CLINICAL TRIAL: NCT02870920
Title: A Phase II Randomized Study of Durvalumab and Tremelimumab and Best Supportive Care vs Best Supportive Care Alone in Patients With Advanced Colorectal Adenocarcinoma Refractory to Standard Therapies
Brief Title: Durvalumab and Tremelimumab and Best Supportive Care vs Best Supportive Care in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO26
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Supportive Care (Active Comparator): Best supportive care available
  Interventions: Other: Best Supportive Care
- Durvalumab plus Tremelimumab and Best Supportive Care (Experimental): Tremelimumab 75mg IV 60 minutes Day 1, cycles 1-4 Durvalumab 1500mg IV 60 minutes Day 1 every 28 days. Plus best supportive care
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Other: Best Supportive Care

INTERVENTIONS:
Drug: Tremelimumab
  Arms: Durvalumab plus Tremelimumab and Best Supportive Care
Drug: Durvalumab
  Other Names: Imfinzi
  Arms: Durvalumab plus Tremelimumab and Best Supportive Care
Other: Best Supportive Care

SUMMARY:
The standard or usual treatment for this disease is treatment with drugs and other treatments that may help to make a patient better or may improve their quality of life. This treatment is known as "best supportive care" (BSC). Although patients with best supportive care can feel better for some months, the cancer usually continues to grow.

DETAILED DESCRIPTION:
Durvalumab is a new type of drug for many types of cancer. Laboratory tests show that it works by allowing the immune system to detect cancer and reactivate the immune response. This may help to slow down the growth of cancer or may cause cancer cells to die. Durvalumab has been shown to shrink tumours in animals and has been studied in a few people and seems promising but it is not clear if it can offer better results than standard treatment alone.

Tremelimumab is a new type of drug for various types of cancers. It works in a similar way to durvalumab and may improve the effect of durvalumab. This may also help slow the growth of the cancer cells or may cause cancer cells to die. Tremelimumab has been shown to shrink tumours in animals and has been studied in a few people and seems promising but it is not clear if it can offer better results than standard treatment alone when used with durvalumab.

Combinations of durvalumab and tremelimumab have also been studied and when combined have been shown to increase tumour shrinkage in animals compared to either drug alone and while the combination has been studied in a few people, it is not clear if it can offer better results than standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or pathologically confirmed advanced (metastatic or locally advanced) colorectal cancer that is unresectable.
* Received a prior thymidylate synthase inhibitor (e.g. 5-fluorouracil (5-FU), capecitabine, raltitrexed, UFT) for metastatic disease or as adjuvant therapy. A thymidylate synthase inhibitor may have been given in combination with oxaliplatin or irinotecan.
* Received and failed an irinotecan -containing regimen (i.e. single-agent or in combination) for treatment of metastatic disease, OR relapsed within 6 months of completion of an irinotecan-containing adjuvant therapy, OR have documented unsuitability for an irinotecan-containing regimen.
* Received and failed an oxaliplatin-containing regimen (i.e. single-agent or in combination) for treatment of metastatic disease, OR relapsed within 6 months of completion of an oxaliplatin-containing adjuvant therapy OR have documented unsuitability for an oxaliplatin-containing regimen.
* For patients with colorectal cancer that is RAS-wild type:

Received and failed a cetuximab or panitumumab-containing regimen (i.e. single-agent or in combination) for treatment of metastatic disease OR have documented unsuitability for a cetuximab or panitumumab-containing regimen

* Patient prior treatment with VEGF targeting therapy, such as bevacizumab, aflibercept, ramucirumab, or regorafenib, is permitted but not mandatory. Reasons not used are to be documented.
* Patient prior treatment with TAS-102 (an agent composed of a combination of trifluorothymidine (FTD) and tipiracil hydrochloride (TPI)), is permitted but not mandatory.
* The only remaining standard available therapy as recommended by the Investigator, in consultation with the patient, is best supportive care.
* Must have presence of measurable or evaluable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST 1.1).
* Imaging investigations including CT/MRI of chest/abdomen/pelvis or other scans as necessary to document all sites of disease done within 28 days prior to randomization.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of ≥ 12 weeks at the time of study entry.
* Must be ≥ 18 years of age.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.
* Patient must consent to provision of, and investigator(s) must confirm adequacy of tissue, and confirm access to and agree to submit within 4 weeks of randomization to the CCTG Central Tumour Bank, a representative formalin fixed paraffin block of tumour tissue in order that the specific correlative marker assays may be conducted.
* Patient must consent to provision of samples of blood in order that the specific correlative marker assays
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French.

Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.

* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient randomization.
* The patient is not receiving therapy in a concurrent clinical study and the patient agrees not to participate in other clinical studies during their participation in this trial while on study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, Study Chair — Univ. Health Network-Princess Margaret Hospital, Toronto ON Canada
Locations (25):
- Canada (25):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - L'Hotel-Dieu de Levis, Lévis, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Centre Integre Universitaire De Sante Et De Services, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen EX, Jonker DJ, Loree JM, Kennecke HF, Berry SR, Couture F, Ahmad CE, Goffin JR, Kavan P, Harb M, Colwell B, Samimi S, Samson B, Abbas T, Aucoin N, Aubin F, Koski SL, Wei AC, Magoski NM, Tu D, O'Callaghan CJ. Effect of Combined Immune Checkpoint Inhibition vs Best Supportive Care Alone in Patients With Advanced Colorectal Cancer: The Canadian Cancer Trials Group CO.26 Study. JAMA Oncol. 2020 Jun 1;6(6):831-838. doi: 10.1001/jamaoncol.2020.0910. PMID 32379280
- [Result] Eric X. Chen, MD, PhD; Jonathan M. Loree, MD; Emma Titmuss, MSc; Derek J. Jonker, MD; Hagen F. Kennecke, MD; Scott Berry, MD; Felix Couture, MD; Chaudharry E. Ahmad, MD; John R. Goffin, MD; Petr Kavan, MD; Mohammed Harb, MD; Bruce Colwell, MD; Setareh Samimi, MD; Benoit Samson, MD; Tahir Abbas,MD; Nathalie Aucoin, MD; Francine Aubin, MD; Sheryl Koski, MD; Alice C.Wei, MD; Dongsheng Tu, PhD; Chris J. O'Callaghan, PhD
- [Derived] Ma LX, Titmuss E, Loree JM, Jonker DJ, Kennecke HF, Berry S, Couture F, Ahmad CE, Goffin JR, Kavan P, Harb M, Colwell B, Samimi S, Samson B, Abbas T, Aucoin N, Aubin F, Koski S, Tu D, O'Callaghan C, Chen EX. Plasma arginine as a predictive biomarker for outcomes with immune checkpoint inhibition in metastatic colorectal cancer: a correlative analysis of the CCTG CO.26 trial. J Immunother Cancer. 2024 Dec 4;12(12):e010094. doi: 10.1136/jitc-2024-010094. PMID 39631846
- [Derived] Topham JT, O'Callaghan CJ, Feilotter H, Kennecke HF, Lee YS, Li W, Banks KC, Quinn K, Renouf DJ, Jonker DJ, Tu D, Chen EX, Loree JM. Circulating Tumor DNA Identifies Diverse Landscape of Acquired Resistance to Anti-Epidermal Growth Factor Receptor Therapy in Metastatic Colorectal Cancer. J Clin Oncol. 2023 Jan 20;41(3):485-496. doi: 10.1200/JCO.22.00364. Epub 2022 Aug 25. PMID 36007218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 10, 2016 to June 29, 2017 in 27 cancer centres in Canada
Groups:
- Best Supportive Care: Best supportive care available
  Best Supportive Care
- Durvalumab Plus Tremelimumab and Best Supportive Care: Tremelimumab 75mg IV 60 minutes Day 1, cycles 1-4 Durvalumab 1500mg IV 60 minutes Day 1 every 28 days. Plus best supportive care
  Tremelimumab
  Durvalumab
  Best Supportive Care
Period: Overall Study
Arm/Group | Best Supportive Care | Durvalumab Plus Tremelimumab and Best Supportive Care
Started | 61 | 119
Completed | 61 | 119
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Best Supportive Care | Durvalumab Plus Tremelimumab and Best Supportive Care | Total
Number analyzed (Participants) | 61 | 119 | 180
Age, Customized [Count of Participants; unit: Participants]
  Younger than 65 years | 31 | 56 | 87
  65 years or older | 30 | 63 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 45 | 59
  Male | 47 | 74 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 3 | 16 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  White | 54 | 97 | 151
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 61 | 119 | 180
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 17 | 33 | 50
    1 | 44 | 86 | 130

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from randomization to death from any cause with patients who were alive at the time of the final analysis or who became lost to follow-up censored at their last date known to be alive.
Time Frame: 24 months
Population: All randomized patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Best Supportive Care | Durvalumab Plus Tremelimumab and Best Supportive Care
Number analyzed (Participants) | 61 | 119
months | 4.1 [3.3 to 6.0] | 6.6 [6.0 to 7.4]
Statistical Analysis 1: Comparison: Best Supportive Care vs Durvalumab Plus Tremelimumab and Best Supportive Care; Test type: Superiority; p = 0.07, Log Rank; Hazard Ratio (HR) = 0.72, 90% CI 2-sided [0.54 to 0.97]

2. Secondary Outcome: Progression-free Survival
Description: Defined as the time from randomization to the first objective documentation of disease progression, defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions, or death due to any cause with patients who had not progressed or died at the time of final analysis censored on the date of the last tumour assessment.
Time Frame: 24 months
Population: All randomized patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Best Supportive Care | Durvalumab Plus Tremelimumab and Best Supportive Care
Number analyzed (Participants) | 61 | 119
Months | 1.9 [1.8 to 1.9] | 1.8 [1.8 to 1.9]
Statistical Analysis 1: Comparison: Best Supportive Care vs Durvalumab Plus Tremelimumab and Best Supportive Care; Test type: Superiority; p = 0.97, Log Rank; Hazard Ratio (HR) = 1.01, 90% CI 2-sided [0.76 to 1.34]

3. Secondary Outcome: Objective Response Rate
Description: Defined as percentage of participants with objective response over all participants randomized. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 24 months
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Best Supportive Care | Durvalumab Plus Tremelimumab and Best Supportive Care
Number analyzed (Participants) | 61 | 119
Participants
  Responded | 0 | 1
  Not responded | 61 | 118

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Best Supportive Care | Durvalumab Plus Tremelimumab and Best Supportive Care
All-Cause Mortality (participants affected / at risk) | 54/61 | 100/118
Serious Adverse Events (participants affected / at risk) | 0/61 | 55/118
Other Adverse Events (participants affected / at risk) | 51/61 | 116/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Best Supportive Care (N=61) | Durvalumab Plus Tremelimumab and Best Supportive Care (N=118)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 2
Colonic obstruction (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 3
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 4
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Other gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 0 | 3
Fatigue (General disorders) | 0 | 2
Fever (General disorders) | 0 | 4
Flu like symptoms (General disorders) | 0 | 1
Other general disorders, administration site conditions (General disorders) | 0 | 1
Other immune system disorders (Immune system disorders) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 0 | 5
Urinary tract infection (Infections and infestations) | 0 | 2
Other infections and infestations (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Intestinal stoma obstruction (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 3
Cardiac troponin T increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 2
Lipase increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Edema cerebral (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | NA | 1
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Best Supportive Care (N=61) | Durvalumab Plus Tremelimumab and Best Supportive Care (N=118)
Hypothyroidism (Endocrine disorders) | 1 | 10
Abdominal distension (Gastrointestinal disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 18 | 53
Constipation (Gastrointestinal disorders) | 14 | 49
Diarrhea (Gastrointestinal disorders) | 6 | 37
Dry mouth (Gastrointestinal disorders) | 2 | 11
Dyspepsia (Gastrointestinal disorders) | 7 | 17
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 17 | 53
Vomiting (Gastrointestinal disorders) | 9 | 30
Other gastrointestinal disorders (Gastrointestinal disorders) | 2 | 10
Chills (General disorders) | 1 | 10
Edema limbs (General disorders) | 12 | 14
Fatigue (General disorders) | 34 | 91
Fever (General disorders) | 6 | 15
Flu like symptoms (General disorders) | 1 | 9
Non-cardiac chest pain (General disorders) | 1 | 6
Pain (General disorders) | 9 | 27
Urinary tract infection (Infections and infestations) | 0 | 14
Weight loss (Investigations) | 1 | 23
Anorexia (Metabolism and nutrition disorders) | 22 | 60
Dehydration (Metabolism and nutrition disorders) | 1 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 10
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 8
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 21
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 | 6
Dizziness (Nervous system disorders) | 1 | 6
Dysgeusia (Nervous system disorders) | 3 | 8
Headache (Nervous system disorders) | 4 | 15
Paresthesia (Nervous system disorders) | 2 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 18 | 40
Anxiety (Psychiatric disorders) | 7 | 13
Confusion (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 11 | 43
Hematuria (Renal and urinary disorders) | 2 | 6
Urinary frequency (Renal and urinary disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 41
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 45
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 23
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 28
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT02870920/Prot_001.pdf
  • Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT02870920/SAP_000.pdf